CLINICAL TRIAL: NCT04860648
Title: The Second Affiliated Hospital of Zhejiang University, School of Medicine
Brief Title: Lung Ultrasound Guided Prevention of Postoperative Pulmonary Complications in Moderate to High Risk Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-0127
Record Dates: First submitted 2021-03-28; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Respiratory Complication
Keywords: lung ultrasound, postoperative pulmonary complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LUS group (Experimental): patients receive lung ultrasound examination, and doctors give the treatment according to the LUS results
  Interventions: Other: lung ultrasound
- Control group (No Intervention): patients receive no lung ultrasound examination and other intervention

INTERVENTIONS:
Other: lung ultrasound — doctors treat the patients combining the Lus results and clinical practice
  Other Names: doctors' clinical decision
  Arms: LUS group

SUMMARY:
Postoperative pulmonary complications (PPCs) occur in many patients, especially those with high risks, and are associated with increased hospital length of stay, morbidity and costs of care. According to European Perioperative Clinical Outcome definitions, major pulmonary complications include atelectasis, respiratory infection, pleural effusion, and pneumothorax. Because identifying patients at high risk for PPCs may allow earlier treatment, predictive scores ( the Assess Respiratory Risk in Surgical Patients in Catalonia score [ARISCAT]) have been developed.Lung ultrasound (LUS) is more accurate than chest X-ray in diagnosing pulmonary complications, and lung ultrasound performed in the postanesthesia care unit may identify patients at higher risk for pulmonary complications. So we aimed to study if lung ultrasound can guide the prevention of PPCs in moderate to high risk patients.

DETAILED DESCRIPTION:
patients recruited are randomized into the two groups: LUS group and Control group. Patients in LUS group received ultrasound examination and guided the treatment according to the ultrasound results, while the control group did not receive ultrasound examination, just the same as the routine clinical practice. This study aims to explore whether ultrasound-guided clinical treatment can reduce the incidence of postoperative pulmonary complications in moderate to highrisk patients. Before operation, informed consent was signed according to the inclusion criteria, and the incidence of pulmonary complications within 5 days after operation (or before discharge) was recorded after operation.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 Estimated ARISCAT score ≥26分

Exclusion Criteria:

* transferred to ward or ICU directly day surgery (patients won't stay in hospital longer than 24 hours after surgery actual ARISCAT score < 26分 the technical incompatibility of the acoustic window patients refused pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
the incidence of postoperative pulmonary complications | within 5 days after operation or before discharge, whichever came first
  postoperative pulmonary complications are defined as a composite outcome including respiratory infection, respiratory failure,pleural effusion, atelectasis,pneumothorax,broncospasm and aspiration pneumonitis

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, MD, Study Chair — Zhejiang University
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China